CLINICAL TRIAL: NCT06308146
Title: Evaluating the Efficacy of Bacillus Subtilis ATCC 122264 on Intestinal Gas Symptoms and Quality of Life in Participants With Functional Bloating: a Randomized, Double-blind, Placebo-controlled, 2-arm Parallel Study
Brief Title: Effect of Bacillus Subtilis ATCC 122264 Supplementation on Gas Symptoms and Quality of Life in Participants With Functional Bloating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kerry Group P.L.C (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S21-1249496
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Functional Bloating

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to receive either the probiotic or placebo. Study products (i.e., TP and placebo) will be dispensed by the site as per the randomization scheme at the study visits.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To minimize bias, the sponsor representatives involved in the study, the investigator, the participants, and any healthcare professionals or site personnel involved in participant management or outcome assessment remained blinded to interventional assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic, Bacillus subtilis (Experimental): Bacillus subtilis ATCC 122264; One capsule per day with a larger meal; providing 5 billion CFU for 8 weeks.
  Interventions: Dietary Supplement: Bacillus subtilis ATCC 122264
- Placebo (Placebo Comparator): Placebo; matched the test product in colour, size, smell and texture and contained only the excipients (maltodextrin and hydroxypropylmethylcellulose); one capsule per day with a larger meal, for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bacillus subtilis ATCC 122264 — One capsule (5 billion CFU) per day for 8 weeks.
  Arms: Probiotic, Bacillus subtilis
Dietary Supplement: Placebo — One capsule per day for 8 weeks.
  Arms: Placebo

SUMMARY:
A randomized, double blind, placebo-controlled, 2-arm parallel study to evaluate the efficacy of Bacillus subtillis in providing relief and improving quality of life in participants suffering from functional abdominal bloating/distension when administered for a period of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult participants who are 18 to 65 years of age (inclusive).
* Have a body mass index (BMI) between 18.5 to 34.9 kg/m2 (inclusive).
* In good general health (no active or uncontrolled diseases or conditions).
* Participants with Functional Abdominal Bloating/Distension, defined by ROME IV criteria as below: Must meet both of the following diagnostic criteria fulfilled for the last three months with symptom onset ≥ 6 months prior to diagnosis: a) Recurrent bloating and/or distension occurring on average at least 1 day/week, and abdominal bloating and/or distension predominates over other symptoms (bloating-related mild pain may be present as well as minor bowel movement abnormalities). b) There are insufficient criteria for a diagnosis of irritable bowel syndrome, functional constipation, functional diarrhea, or post-prandial distress syndrome.
* Individuals of childbearing potential must have negative urine pregnancy result at baseline and agree to practice acceptable form of birth control for a certain period prior to the first dose of study product and throughout the study duration.
* Individuals with the potential to get others pregnant must agree to use condom or other acceptable methods to prevent pregnancy throughout the study. Complete abstinence from sexual intercourse that can result in pregnancy is also acceptable.
* Be willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, carry out all study-related procedures, communicate effectively with the study staff, and agree to allow evaluations related to digestive health.
* Agree to refrain from treatments in the defined timeframe, as outlined in the protocol.
* Agree not to change current dietary habits known to alter GI function (including, but not limited to, iron supplements) within the 4 weeks prior to baseline visit or anytime during the study duration.
* Agree not to change smoking and alcohol consumption habits, and activity/training levels two weeks prior to baseline and for the duration of the study.

Exclusion Criteria:

* Individuals who are lactating, pregnant or planning to become pregnant during the study duration.
* Have a known sensitivity, intolerability, or allergy to wheat, soy or milk or any other ingredients of the study products or their excipients, or all of the rescue medications as outlined in the protocol.
* An unexplained weight loss of ≥5% of body weight in one month or ≥10% over a period of six months as assessed at screening.
* Received a vaccine for COVID-19 in the 2 weeks prior to screening or during the study period, current COVID-19 infections, or currently have the post COVID-19 condition as defined by World Health Organization (WHO) (i.e., individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis).
* Known medical history of organic disease including IBS, inflammatory bowel disease (IBD; including ulcerative colitis and Crohn's disease), functional constipation and diarrhea (defined by the Rome IV diagnostic criteria), celiac disease, gluten intolerance/sensitivity, a benign or malignant tumor of intestine or colon or significant systemic disease, self-reported lactose intolerance and/or malabsorption, gastroparesis, gastroenteritis, endometriosis, diverticulosis, gastric or duodenal ulcers, history of intestinal surgery (excluding appendectomy or herniorrhaphy), history of bariatric surgery, pancreatitis, or eating disorder.
* Major surgery in the past 3 months or individuals who have planned surgery during the course of the study, or participants who have had a colonoscopy in past 3 months.
* Use of concomitant treatments within the defined timeframe, as outlined in the protocol.
* Change from current routine/ standard dietary habits (e.g., newly starting or modifying current restrictive diet such as FODMAP diet, ketogenic diet, vegan diet etc. or notable change in eating habits e.g., significant change in number of daily meals) within the 4 weeks prior to the baseline visit or anytime during the study duration.
* Having a history of heart disease, uncontrolled high blood pressure (≥140 systolic or

  * 90 diastolic mmHg), renal or hepatic impairment/disease, uncontrolled diabetes (Type I or Type II), bipolar disorder, hepatic or renal dysfunction, unstable thyroid disease, immune disorders and/or immunocompromised (e.g. HIV/AIDS), a history of cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit), or a history of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential participant at risk because of participation in the study, or influence the results or the potential participant's ability to participate in the study.
* History of alcohol or substance abuse in the 12 months prior to screening (including having been hospitalized for such in an in-patient or out-patient intervention program).
* Receipt or use of test product(s) in another research study within 30 days prior to the baseline visit.
* Any other active or unstable medical conditions or use of medications/supplements/ therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant or the quality of the study data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-10-11 (Actual); Study Completion 2022-10-11 (Actual)

PRIMARY OUTCOMES:
Effect on intestinal gas symptoms and quality of life | 8 weeks
  to evaluate change from baseline in IGQ score at Week 8 between groups. The Intestinal Gas Questionnaire (IGQ) is a 17-item questionnaire that assesses the severity of six GI-related symptoms and their impact on the quality of life. The global score is between (0-100) with higher score means worst symptoms or impact.

SECONDARY OUTCOMES:
Effect on intestinal gas symptoms and quality of life | 4 weeks
  to evaluate change from baseline in IGQ score at Week 4 between groups The Intestinal Gas Questionnaire (IGQ) is a 17-item questionnaire that assesses the severity of six GI-related symptoms and their impact on the quality of life. The global score is between (0-100) with higher score means worst symptoms or impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Apex Trials, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] LeMoire A, Lin L, Girard SA, Baisley J, Wang J, Atif A, Zahra R, Millette M. Effect of Bacillus subtilis ATCC 122264 on intestinal gas symptoms and quality of life in adults with functional bloating. Benef Microbes. 2025 Jan 28;16(3):281-292. doi: 10.1163/18762891-bja00057. PMID 39929203